CLINICAL TRIAL: NCT01626183
Title: Molecular Taxonomy in Pediatric Cancer- IncRNA Expression in Primary T-ALL
Brief Title: Studying RNA in Samples From Younger Patients With T-Cell Acute Lymphoblastic Leukemia
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: AALL12B8; COG-AALL12B8 (Other: Children's Oncology Group); CDR0000735509 (Other: clinicaltrials.gov); NCI-2012-01980 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-06-20; First posted 2012-06-22 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Leukemia
Keywords: T-cell childhood acute lymphoblastic leukemia; recurrent childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — RNA
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: RNA analysis
Genetic: proteomic profiling
Other: laboratory biomarker analysis

SUMMARY:
RATIONALE: Studying samples of blood and tissue from patients with cancer in the laboratory may help doctors identify and learn more about biomarkers related to cancer

PURPOSE: This laboratory study is looking into RNA in samples from younger patients with T-cell (T) acute lymphoblastic leukemia (ALL).

DETAILED DESCRIPTION:
OBJECTIVES:

* Characterization of the transcriptomic landscape in diagnosis and relapse of T-cell acute lymphoblastic leukemia (ALL) and the direct comparison with corresponding physiological samples (human thymus).
* Perform high-throughput transcriptome ribonucleic acid (RNA) sequencing using matched diagnostic T-precursor pediatric ALL samples (peripheral blood or bone marrow).

OUTLINE: Archived peripheral blood and bone marrow samples are analyzed for long non-coding RNA (IncRNA) expression and sequencing.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Peripheral blood and bone marrow samples from pediatric patients with diagnosed and relapsed T-ALL

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pediatric patients with diagnosed or relapsed T-ALL
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Identification and characterization of IncRNA of pediatric T-cell acute lymphoblastic leukemia

CONTACTS AND LOCATIONS:
Overall Officials: Iannis Aifantis, PhD, Principal Investigator — NYU Langone Health